CLINICAL TRIAL: NCT00949936
Title: Debilitating Low Back paIn: Multi-centre Safety and performanCe invEstigation Of CAdiscTM-L, Total Disc ReplacemeNt Therapy
Brief Title: Safety and Performance Study of the CAdiscTM-L Lumbar Spinal Disc Replacement Device For CE Marking
Acronym: DISCERN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranier Technology Limited (Industry)
Responsible Party: Ian Quirk : Worldwide Clinical & Regulatory Affairs Director, Ranier Technology Ltd
Purpose: Treatment
Other Study IDs: Ranier01/2008
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Chronic Low Back Pain; Lumbar Degenerative Disc Disease
Keywords: Spine surgery
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Total Disc Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: CAdisc™-L (Total Disc Replacement)

SUMMARY:
The purpose of this European Union (EU) study to evaluate the safety and performance of the CAdiscTM-L Lumbar Spinal Disc Replacement Device in the surgical replacement of the lumbar intervertebral discs (L3 to S1) for patients requiring surgical intervention for total lumbar disc replacement for the treatment of debilitating, chronic low back pain.

DETAILED DESCRIPTION:
Study Design: International, multicenter, open, clinical investigation with comparison to pre-operative

Currently there are two surgical procedures for the treatment of chronic low back pain: Spinal fusion and Total Disc Replacement. CAdisc™-L(Compliant Artificial disc - Lumbar) is a Lumbar total disc replacement product that preserves motion and restores disc height and stability

Surgical access is via a routine anterior approach with discectomy (removal of the diseased disc), which is performed prior to implantation of the CAdisc™-L. Instruments are then used to prepare the disc space and to controllably place the replacement disc at the target point. It is not intended for the surgery to differ in type, duration or risk to any other device of this nature.

ELIGIBILITY:
Inclusion Criteria:

* Male or non pregnant, non-lactating female
* Aged between 25-65 years (inclusive)
* BMI < 35
* Preoperative ODI > 30 points
* Chronic low back pain, and is in the opinion of the investigator a suitable candidate for anterior lumbar surgery
* Completed at least 6 months of conservative treatment without obtaining adequate symptomatic relief
* Degenerative disc changes at a single level between L3 - L4, or L4 - L5, or L5 - S1 as confirmed by positive discography and visualized by X-Ray, CT or MRI scan and/or with one or more of the following:

  * Decrease in disc height < 50% (or up to 80% and no benefit from facet injections)
  * Annular thickening
  * Herniated nucleus pulpous
* Subject is able to give voluntary, written informed consent to participate in this investigation and from whom written consent must be obtained prior to enrolment.

Exclusion Criteria:

* Back or leg pain of unknown aetiology
* Radicular or sciatic pain which is more severe than low back pain
* Previous lumbar spinal surgery which could affect the trial outcome (e.g., disc replacement)
* Obvious signs of psychological or worker's compensation or litigation claim elements to their condition, or are actively engaged in such activities
* Subject is unwilling or unable to give consent or adhere to the follow-up programme
* Active infection or metastatic disease
* Non-degenerative spondylolisthesis
* Degenerative spondylolisthesis > grade 1
* Known allergy to any of the implant materials
* Osteoporosis (if suspected to be confirmed by bone density being 2.5SD below normal as assessed using DEXA analysis in post-menopausal females if suggested by X-ray or other risk factors)
* Osteopenia
* Bony lumbar stenosis
* Pars defect
* Isolated radicular compression syndromes, especially due to disc herniation
* Clinically compromised vertebral bodies at the affected levels due to current or past trauma
* Subject is skeletally immature as determined by the investigator
* Subject has participated in another clinical investigation or study with an investigational medical device within the last 60 days
* Concomitant medications that are known significantly to interfere with bone/soft tissue healing, e.g. steroids.
* Uncorrected iliac, aorto-iliac, or aortic aneurysm disease.
* Spinal instability (> 3mm translation or > 5° angulation) confirmed by functional radiological assessment.
* Degenerative disc changes at the L6 - S1 level

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2009-10; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Improvement of 15 points on the Oswestry Disability Index (ODI) scale at 3 months post-surgery, compared to baseline

CONTACTS AND LOCATIONS:
Locations (4):
- Antwerp, Belgium
- Bogen, Germany
- Zwolle, Netherlands
- Aberdeen, United Kingdom